CLINICAL TRIAL: NCT02289781
Title: Wear of Enamel Antagonists by Polished Ceramic Surfaces
Brief Title: Wear of Enamel Against Polished Zirconia Crowns
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: 3M Pharmaceuticals Pty Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201200002; 00104254 (Other Grant/Funding Number: 3M ESPE)
Record Dates: First submitted 2014-11-07; First posted 2014-11-13 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Tooth Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Zirconia posterior crowns: Monolithic zirconia crowns which are polished and non-glazed
  Interventions: Device: posterior crowns
- Metal-Ceramic posterior crowns: Metal-supported glass-ceramic veneered crowns which are polished and non-glazed
  Interventions: Device: posterior crowns

INTERVENTIONS:
Device: posterior crowns — teeth will be prepared to receive posterior crown made of either zirconia or metal-ceramic material

SUMMARY:
A randomized, controlled clinical trial is designed to analyze the wear of enamel by opposing polished monolithic zirconia crowns and by the polished veneer surfaces of metal-ceramic crowns. This single-blind pilot study will involve a total of 30 teeth that require full coverage crowns that oppose natural antagonist teeth.

The objectives of this research are to test the following hypotheses: (1) differences between mean wear of antagonist enamel by polished monolithic zirconia crowns and by the polished veneer surface of metal-ceramic crowns are statistically significant; (2) differences between mean wear of antagonist enamel by opposing polished monolithic zirconia crowns and enamel by opposing enamel are statistically significant; and (3) differences between mean antagonist wear of enamel by opposing polished veneer surfaces of metal-ceramic crowns and enamel by opposing enamel are statistically significant.

DETAILED DESCRIPTION:
To participate in this study a crown will need to be place on one of the back teeth. This generally occurs when the back tooth has a big filling and there is a risk for fracture of the tooth or a root canal has been performed on the tooth. An initial x-ray of the tooth and the surrounding teeth will be done to make sure that there is enough bone supporting the tooth that will be crowned.

A receive local anesthesia will be used in the area where the crown will be made. The tooth area may need to be build-up with a filling material if there is not enough tooth structure remaining. Once this happens, then a high-speed drill will be used to a grind down of the tooth material using to a make smaller size of the original tooth. A small thread will be used to make space between the gums and tooth so an accurate replica of the tooth can be made. A temporary crown will be made to go over the prepared tooth and will cement until the final crown is ready to be cemented.

The extra procedures will be done to measure bite force to see how much force is exerted with the teeth. Other extra procedures include the six month and yearly impressions as well as scanning of your teeth to aid in the measurement of wear.

Participants will be randomly assigned (much like the flip of a coin) to receive either a crown that has metal in it or a crown that is all-ceramic. Both of these materials are considered standard of care in dental practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be over 21 years of age and in good overall health. No contraindications to dental treatment are present
* Subjects must be in good overall good dental health and are at a low caries risk, with no active tooth decay (caries), and no periodontal disease. Periodontal pocket depths on all remaining teeth are not greater than 4 mm
* Subjects must have no existing temporomandibular disorder, (e.g. clicking, popping, pain on opening) or parafunctional habits (e.g. bruxism, clenching)
* Subjects must need a crown on either a first or second premolar or first or second molar in any arch. Abutment teeth must be restorable and have a crown:root ratio of at least 1:1. Abutment teeth must have a full complement of opposing non-restored or minimally restored natural teeth. Minimally restored means the teeth contain no restoration greater than a Class II amalgam restoration. The opposing arch must not have a full coverage restoration or a partial denture. The contralateral tooth and its antagonist are present
* Subjects must exhibit good oral hygiene and compliance with oral hygiene instructions as determined by the amount of plaque present on tooth surfaces
* Subjects must exhibit a normal flow of saliva. Subjects with any medical pathologies that limit salivary flow volume or who require a chronic intake of medications that minimize flow of saliva will be excluded from the study
* Subjects must be willing to pay $500 for the clinic incidentals and they must be compliant with yearly appointments

Exclusion Criteria:

* anything that does not meet inclusion criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients accessing care in a dental clinc needing full coverage crowns.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline, 1 year, 2 years, and 3 years wear of Enamel Antagonist | Change from baseline, 1 year, 2 years, and 3 years
  The wear of the enamel opposing the monolithic zirconia will be measured and compared with wear with the metal-ceramic crowns by using scanning technology to scan the teeth at baseline and then at the succeeding time periods. Also, impressions of the teeth will be used on a laser scanner to measure the volume loss on the crowns and the opposing teeth.

SECONDARY OUTCOMES:
Change from baseline, 1 year, 2 years, and 3 years in the wear of Zirconia and Metal-Ceramic Crowns | Change from baseline, 1 year, 2 years, and 3 years
  The wear of the enamel opposing the monolithic zirconia will be measured and compared with wear with the metal-ceramic crowns by using scanning technology to scan the teeth at baseline and then at the succeeding time periods. Also, impressions of the teeth will be used on a laser scanner to measure the volume loss on the crowns and the opposing teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine F. Esquivel-Upshaw, D.M.D., M.S., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] F Esquivel-Upshaw J, Hsu SM, Bohorquez AC, Abdulhameed N, Scheiffele GW, Kim M, Neal D, Chai J, Ren F. Novel methodology for measuring intraoral wear in enamel and dental restorative materials. Clin Exp Dent Res. 2020 Dec;6(6):677-685. doi: 10.1002/cre2.322. Epub 2020 Sep 21. PMID 32955159